CLINICAL TRIAL: NCT04993144
Title: To Explore the Therapeutic Effects of Continuous Theta-burst Stimulation Over Left Dorsolateral Prefrontal Cortex in Autism Spectrum Disorder
Brief Title: The Therapeutic Effects of Continuous Theta Burst Stimulation in Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201802246A0
Record Dates: First submitted 2021-07-12; First posted 2021-08-06 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active (Active Comparator): Participants received the real intervention of TBS (cTBS 600) over the left dorsolateral prefrontal cortex for 8 weeks (2 days/week).
  *cTBS = continuous theta burst stimulation
  Interventions: Device: continuous theta burst stimulation
- Sham (Sham Comparator): Participants received the sham intervention of TBS (coil tilted one-wing 90° off the head) over the left dorsolateral prefrontal cortex for 8 weeks (2 days/week).
  Interventions: Device: continuous theta burst stimulation
- Normal control (No Intervention): No intervention.

INTERVENTIONS:
Device: continuous theta burst stimulation — stimulatory protocol
  Arms: Active; Sham

SUMMARY:
The investigator would like to investigate the impact of theta burst stimulation over left dorsolateral prefrontal cortex in autism spectrum disorder

ELIGIBILITY:
Inclusion Criteria:

* autism spectrum disorder, confirmed by ADOS

Exclusion Criteria:

* current and past systemic disease
* current and past major psychiatric disorders including schizophrenia, bipolar affective disorder and major depressive disorder
* current and past brain injuries
* intelligence < 70
* seizure history
* pregnant

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Changes of total scores of Social Responsiveness Scale | baseline; post TBS (8 weeks after baseline); One month follow up (4 weeks after post TBS)
  Social Responsiveness Scale can measure the autism clinical severity with the range from 65-260. The lower scores stand for better social responsiveness.
Changes of total scores of Repetitive Behavior Scale-Revised | baseline; post TBS (8 weeks after baseline); One month follow up (4 weeks after post TBS)
  Repetitive Behavior Scale-Revised is a questionnaire that focuses on repetitive behavior. The score ranges from 0-129. The lower scores stand for lower repetitive behavior.

SECONDARY OUTCOMES:
Changes of total scores of Emotional Dysregulation Inventory | baseline; post TBS (8 weeks after baseline); One month follow up (4 weeks after post TBS)
  Emotional Dysregulation Inventory is a parents' report questionnaire for emotional dysregulation. The score ranges from 0-120. The lower scores stand for better emotional regulation.
Changes of total scores of Adaptive Behavior Assessment System | baseline; post TBS (8 weeks after baseline); One month follow up (4 weeks after post TBS)
  Adaptive Behavior Assessment System is a parents' report questionnaire for adaptive behavior. The score ranges from 9-171. The higher scores stand for better adaptive behavior.
Changes of total scores of Vineland Adaptive Behavior Scales | baseline; post TBS (8 weeks after baseline); One month follow up (4 weeks after post TBS)
  Vineland Adaptive Behavior Scales is a parents' report questionnaire for adaptive behavior. The score ranges from 0-484. The higher scores stand for better adaptive behavior.
Changes in accuracy of Frith-Happe animation | baseline; post TBS (8 weeks after baseline); One month follow up (4 weeks after post TBS)
  A quick and objective test of Theory of Mind. 8 questions in total, the more correct questions stand for better Social Cognition.
Changes in accuracy of Eyes task | baseline; post TBS (8 weeks after baseline); One month follow up (4 weeks after post TBS)
  An advanced test for Theory of Mind. 43 questions in total, the more correct questions stand for better social skills.
Changes in accuracy of Wisconsin Card Sorting Test | baseline; post TBS (8 weeks after baseline); One month follow up (4 weeks after post TBS)
  An advanced test for cognitive flexibility. 128 questions in total, the more correct questions stand for better cognitive flexibility.
Changes of total scores of Behavior Rating Inventory of Executive Function | baseline; post TBS (8 weeks after baseline); One month follow up (4 weeks after post TBS)
  Behavior Rating Inventory of Executive Function is a parents' report questionnaire for executive function. The score ranges from 86-258. The lower scores stand for better executive function.
Raven's Progressive Matrices | baseline; post TBS (8 weeks after baseline); One month follow up (4 weeks after post TBS)
  An advanced test for for executive function. 60 questions in total, the more correct questions stand for better executive function.
Autism Diagnostic Observation Schedule - Generic | baseline; post TBS (8 weeks after baseline)
  The Autism Diagnostic Observation Schedule is a semi-structured assessment of communication, social interaction, and play (or imaginative use of materials) for individuals suspected of having autism spectrum disorders. The social affect domain includes the social and communication items ranging from 0 to 20. The higher scores stand for more clinical severity of autism spectrum disorder.
MRI T1 | baseline; post TBS (8 weeks after baseline)
  Brain structural volumes (cm²)
functional MRI (resting-state/biological motion task) - BOLD signal | baseline; post TBS (8 weeks after baseline)
  Blood-oxygen-level-dependent (BOLD) signal is a measurement used in fMRI, which reflects the neural activity.
Diffusion Tensor Imaging (DTI) - FA | baseline; post TBS (8 weeks after baseline)
  Fractional anisotropy (FA) is a measurement used in DTI, which reflects the movement of water molecules. FA ranges from 0 to 1, the higher FA value may represent more intact axons.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided